# **COVER PAGE**

Date- 04-12-2015. ETHICAL APPROVAL.

Study Title-

Comparative clinical evaluation of coronally advanced flap with

platelet-rich fibrin membrane and chorion membrane in the

treatment of human gingival recession

# MAHATMA JYOTIBA PHULE ROHILKHAND UNIVERSITY, BAREILLY



"COMPARATIVE CLINICAL EVALUATION OF CORONALLY ADVANCED FLAP WITH PLATELET RICH FIBRIN MEMBRANE OR CHORION MEMBRANE IN THE TREATMENT OF HUMAN GINGIVAL RECESSION"

BY

### Dr. BIMMI TRIPATHI

Dissertation Submitted to the Mahatma Jyotiba Phule Rohilkhand University, Bareilly In partial fulfillment of the requirements for the degree of

#### MASTER OF DENTAL SURGERY

In

#### PERIODONTOLOGY AND IMPLANTOLOGY

Year - 2014-2017

Under the Guidance of **Dr. JAISHREE GARG**Reader





# INSTITUTE OF DENTAL SCIENCES

Pilibhit By Pass Road, Bareilly. (U.P.) 243006 INDIA Phone: 0581-2526244 (Reception), 2526051 (Office) Website: www.idsbareilly.in, e-mail: info@idsbareilly.in

#### ETHICAL CLEARANCE CERTIFICATE

To

Dr. Bimmi Tripathi

Post Graduate Student

Department of Periodontology

Institute of Dental Sciences

Bareilly-2430306,

Uttar Pradesh, India

The Institutional Ethical Committee, Institute of Dental Sciences, Bareilly (IDS) has reviewed and discussed your application to conduct the "Interventional Clinical Trial" in the Department of Periodontology, IDS. Your proposal now deemed to meet the requirements of the Institutional Ethical guidelines.

| Approval No. | IDS/ETHCC/14/08 |
|---|---|
| Research Title | Comparative clinical evaluation of coronally advanced flap with platelet rich fibrin membrane and chorion membrane in the treatment of human gingival recession. |
| Approval Date | 04 December 2015 |
| Decision | Approved |

#### Conditions of this approval:

1) The conduct of research should be strictly in accordance with the approved proposal.

2) Report Serious Adverse Event or any other issues related to the research project immediately to the IEC-IDS.

Prof. (Dr.) Sathyajith Naik N.
Principal

Prof. (Dr.) Sathyajith Naik N.

Principal

Institute of Dental Sciences, Bareilly

PATRONAGE

**ROHILKHAND EDUCATIONAL CHARITABLE TRUST** 

## **ABSTRACT**

<u>Background</u>: Platelet-rich fibrin (PRF) is a second-generation platelet concentrate and has the potential to accelerate soft and hard tissue regeneration. The chorion membrane is a fetal tissue. It has been used for its exceptional wound-modulating properties. The aim of the present study was to evaluate and compare the clinical outcome of PRF and chorion membrane in the treatment of isolated Miller's class I or II gingival recession defects.

Materials and methods: A total of 50 recession defects were treated randomly with coronally advanced flap (CAF) along with PRF membrane (site A, n = 25 defects) or CAF with chorion membrane (site B, n = 25 defects). Clinical parameters measured at baseline, 1 month, 3 months and 6 months were recession depth (RD), recession width (RW), clinical attachment level (CAL), width of keratinised gingiva (WKG), plaque index (PI), gingival index (GI) and assessment of gingival biotype. Statistical analysis was performed to compare the treatment outcomes at the follow-up intervals.

Results: Six months after the surgery, statistically significant improvements in mean root coverage, RD, RW, CAL, WKT, PI and GI were observed in both groups. No statistically significant difference was found between the two groups for all of these parameters. The mean percentage of root coverage was  $86.76 \pm 13.76$  in the PRF group (site A) and  $82.89 \pm 15.65$  in the chorion group (site B) at six months post-operatively, with no statistically significant difference between them. The gingival biotype also showed a thick biotype in sites that had an initial thin biotype.

<u>Conclusion</u>: Both PRF and chorion membrane are adequate and predictable treatment modalities for the management of isolated recessed-type defects. Longitudinal studies are needed to confirm these findings.

<u>Keywords</u>: Coronally advanced flap, gingival recession defect, platelet-rich fibrin, root coverage, chorion membrane.

# **Statistical Analysis**

Statistical analysis of the data was done using the statistical package for the social science (SPSS 22.0). The data was compiled using Microsoft excel sheet (windows 2007). For each variable the mean and standard deviation were calculated. The differences between the means were calculated using the Student's paired and independent t-test. p < 0.05 was considered statistically significant.

### Student's t-test:

When sample size is small, 't' test is used to test the hypothesis. This test was designed by **W. S. Gossett**, whose pen name was '**Student**'. Hence this test is also called 'Student's t-test'.

t = ratio of observed difference between two means of small samples to the standard error of difference in the same.

It is applied to find the significance of difference between two proportions as,

- 1. Unpaired 't' test
- 2. Paired 't' test

#### Criteria for applying 't' test,

- 1. The sample must be randomly selected.
- 2. The data must be quantitative.
- 3. The variable is assumed to follow a normal distribution in the population.
- 4. Sample should be less than 30.

## Unpaired (independent) 't' test:

This test is applied to unpaired data of independent observations made on individuals of two different or separate groups or samples drawn from two populations, to test if the difference between the means is real or it can be attributed to sampling variability.

#### Steps:

- As per the null hypothesis, assume that there is no real difference between the means of two samples.
- 2. Find the observed difference between means of two samples  $(\overline{X}_1 \overline{X}_2)$
- 3. Calculate the standard error of difference between the two means.

4. Calculate the 't' value

$$t = \frac{X_1^2 - X_2^2}{SE}$$

5. Determine the pooled degrees of freedom from the formula

$$d.f. = (n_1 - 1) + (n_2 - 1) = n_1 + n_2 - 2$$

6. Compare calculated value with the table value (table of 't') at particular degrees of freedom to find the level of significance.

# Paired "t" test:

It is applied to paired data of independent observations from one sample only when each individual gives a pair of observations.

#### Steps:

- As per the null hypothesis, assume that there is no real difference between the means of two samples.
- 2. Find the difference in each set of paired observations before and after  $(X_1-X_2=X) \label{eq:continuous}$
- 3. Calculate the mean of the differences  $(\overline{X})$
- 4. Work out the standard error of mean, SE = SD/ $\sqrt{n}$
- 5. Determine 't' value

Standard error of difference

- 6. Find the degrees of freedom (n-1)
- Refer 't' table and find the probability of 't' corresponding to n- 1 degree of freedom.
- If the probability is more than 0.05, the difference observed has no significance, because it can be due to chance.

# ANNEXURE – II

# **INFORMED CONSENT**

| Subject: |
|---|
| I, Mr./Mrs./Ms, hereby state that my |
| doctor has provided me with complete details about the proposed procedure/treatment. I have |
| been informed about the purpose of the procedure and the possible risks/complications |
| involved. |
| "I hereby declare that I am fully agreeing, of my own free will, to undergo this procedure/treatment for its successful completion." |
| Patient's Signature: |

# ANNEXURE – III

# DEPARTMENT OF PERIODONTICS & IMPLANTOLOGY INSTITUTE OF DENTAL SCIENCES, BAREILLY (UP)

#### PROFORMA FOR DISSERTATION

| Name: | O.P.D. No: | Date: |
|-------------------------|-------------|-------|
| Address: | Occupation: | Age: |
| | | Sex: |
| CHIEF COMPLAINT: | | |
| PRESENT DENTAL HISTORY: | | |
| PAST DENTAL HISTORY: | | |
| PAST MEDICAL HISTORY: | | |
| PERSONAL HISTORY: | | |
| ORAL HYGIENE HABITS: | | |

| EXAMINATION: GINGIVA: | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| GINGIVAL | WID? | гн: | | | | | | | | | | |
| GINGIVAL | THIC | KNES | SS: | | | | | | | | | |
| RECESSIO | N WII | OTH: | | | | | | | | | | |
| RECESSIO | N DEI | TH: | | | | | | | | | | |
| CLINICAL | ATTA | CHM | ENT I | LEVEI | L: | | | | | | | |
| % OF ROO | T COV | /ERA | GE: (b | aseline | e RD - | RD a | t 1, 3 c | or 6 me | onths) | /baseli | ne RD | ). |
| INDICES: Plaque index (PI): (Silness & Löe, 1967) | | | | | | | | | | | | |
| 17 16 | 15 | 14 | 13 | 12 | 11 | 21 | 22 | 23 | 24 | 25 | 26 | 27 |
| 47 46 | 45 | 44 | 43 | 42 | 41 | 31 | 32 | 33 | 34 | 35 | 36 | 37 |
| Plaque score per tooth =Sum of plaque score on all four surfaces / 4 Total plaque score for a person = Plaque score per tooth / number of teeth examined | | | | | | | | | | | | |

Gingival Index (GI): (Löe and Silness, 1963)

| 17 | 16 | 15 | 14 | 13 | 12 | 11 | 21 | 22 | 23 | 24 | 25 | 26 | 27 |
|----|----|----|----|----|----|----|----|----|----|----|----|----|----|
| 47 | 46 | 45 | 44 | 43 | 42 | 41 | 31 | 32 | 33 | 34 | 35 | 36 | 37 |

| GI Score for the tooth = sum of 4 areas of tooth / 4 |
|------------------------------------------------------|

GI Score for the individual = total indices for each tooth / total no. of teeth examined

#### Clinical Attachment Level (CAL):



| PROVISIONAL DIAGNOSIS:- |
|-------------------------|
| PROGNOSIS:- |
| OVER ALL:- |
| INDIVIDUAL:- |
| INVESTIGATIONS:- |
| FINAL DIAGNOSIS:- |
| TREATMENT PLAN:- |
| CASE SUMMARY: |